CLINICAL TRIAL: NCT05242198
Title: THE EFFECT OF ULTRASOUND GUIDED RECTUS SHEATH BLOCK ON POSTOPERATIVE ANALGESIA AND URETHRAL CATHETER PAIN IN ROBOTIC PROSTATECTOMY OPERATIONS: A PROSPECTIVE RANDOMIZED CONTROLLED TRIAL
Brief Title: Rectus Sheath Block May Relieve Urethral Catheter Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: V.K.V. American Hospital, Istanbul (Other)
Responsible Party: Principal Investigator, Sami Kaan Coşarcan, Dr, V.K.V. American Hospital, Istanbul
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Other
Other Study IDs: Cosarcan2
Record Dates: First submitted 2022-02-07; First posted 2022-02-16 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Prostatectomy
Keywords: regional anesthesia; robotic prostatectomy; fascial plane blocks; postoperative pain; urethral catheter pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rectus sheath block group (Group R) (Other): Patients who underwent rectus sheath block
  Interventions: Procedure: Robotic prostatectomy
- Control group (Group C) (Other): The patients that did not apply any fascial plane block
  Interventions: Procedure: Robotic prostatectomy

INTERVENTIONS:
Procedure: Robotic prostatectomy — patients who will undergo robotic prostatectomy

SUMMARY:
This study aimed to investigate the analgesic efficacy of rectus sheath block and its effect on urethral catheter discomfort in robotic prostatectomy operations.

DETAILED DESCRIPTION:
Our study will be performed on patients who will undergo elective robotic prostatectomy at the American Hospital and Koc University Hospital.All patients will be sedated with midazolam (0.02 mg/kg), following appropriate ASA monitoring and administration of oxygen by mask. All patients will be operated on under general anesthesia. Propofol (Propofol-Lipuro 10mg/ml, Braun) (2 mg/kg), fentanyl (Talinat 0.5mg, Vem İlaç) (0.8µg/kg) and rocuronium (Esmeron 10mg/ml) for the induction of general anesthesia following appropriate monitoring. Following the administration of MSD) (0.6 mg/kg), endotracheal intubation will be performed. For the maintenance of anesthesia, desflurane (Suprane, Baxter) (1 MAC) and remifentanil (Rentanil 2mg, Vem İlaç) (0.05 - 0.2 µg/kg/min) will be administered. Invasive monitoring will be performed on all patients through the radial artery cannula. Depth of anesthesia will be monitored with BIS (Bispectral Index Monitor), and BIS values will be adjusted to be 40-60. In all patients, dexamethasone (Onadron 8mg/2ml, İbrahim Etem) (4mg), ibuprofen 800mg (Intrafen 400mg, Gen İlaç) immediately after intubation and intravenous Paracetamol 1000mg (Parol, Atabay Kimya Sanayi) and Tramadol before extubation to contribute to postoperative analgesia 100 mg (Contramal, Abdi İbrahim İlaç Sanayi) will be administered. In addition, ondansetron (Zofer 4mg, Adeka) (4mg) will be administered for postoperative nausea and vomiting (PONV) prophylaxis.

A rectus sheath block will be applied to one group by randomization in the computer environment, and a fascial plane block will be applied to the other group. At the end of the operation, the anesthesiologist was dressed sterile before the extubation. Surgical drapes and blocks were applied in the supine position without disturbing the sterile environment. Ultrasound and liner probe was covered with a sterile drape. Rectus block, wide bandwidth, high-frequency linear probe (4-12 Mhz) (GE, LOGIQ P9 R3, Seongnam-si, Republic of Korea) and 22 Gauge, 80 mm, insulated facet needle (Pajunk GmbH, Geisingen, Germany) ) was planned. For the rectus sheath block (RB), the ultrasound probe is placed transversely at the level of the umbilicus. The rectus abdominis muscle and fascia transversalis are displayed. The needle is placed on the ultrasound probe from the lateral to the medial by in-plane technique and placed between the posterior sheath of the rectus muscle and the fascia transversalis. 20 ml of 0.25% Bupivacaine plaine (MArcaine, Sanofi İlaç A.Ş, Turkey) is administered after the fascial spread is observed under the rectus abdominis muscle using the hydro dissection technique with saline. For RB, the same procedure is applied to the other parties.

After the patients are extubated, they will be taken to the recovery unit and followed up at 0,10,30, and 60 minutes in pain scores, nausea, vomiting, and other side effects. The pain scores (postoperative pain and urethral catheter-related pain) of the patients transferred from the recovery unit to the service floor will be recorded at the 3rd hour, 6th hour, 12th hour, and 24th hour. To contribute to multimodal analgesia in service follow-ups, intravenous Paracetamol 1000 mg (Parol, Atabay Kimya Sanayi) 3*1 and ibuprofen (Intrafen 400mg, Gene İlaç) 2x400mg will be administered.

Recovery unit (PACU) follow-up; Pain scores of all patients will be recorded at 0, 30, and 60 minutes by blind nurses for the study groups. Patients with NRS scores ≥ 4 will receive 25 µg of fentanyl. Patients with NRS scores ≥ 7 will receive 50 µg of fentanyl. Once NRS scores continue as indicated, fentanyl will be repeated at the same dose at relevant times. The total fentanyl dose requirement in the PACU will be recorded. The PACU unit will record side effects such as nausea, difficulty breathing, and tremors. Urethral catheter pain will also be questioned and recorded at the relevant specified times in the PACU unit. Intravenous morphine patient-controlled analgesia (PCA) will be started in all patients. PCA doses will be adjusted for all patients with only a bolus dose of 1 mg with a 7 min lock time. PCA bolus dose used during the PACU period will be recorded. Patients will be given pain score information for PCA use and instructed to press the bolus button if their pain is four or more.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 - 79, the patients who will undergo robotic prostatectomy surgeries

Exclusion Criteria:

* Presence of a condition preventing facial plane nerve block
* Coagulopathies
* Chronic opioid use
* Stroke
* Polyneuropathy
* Patients with cognitive dysfunction
* Communication difficulties
* Alzheimer's
* Dementia
* Patients who are allergic to the drugs to be used

Ages: 18 Years to 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate operations are specific to the male gender only.
Enrollment: 60 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-09-21 (Actual)

PRIMARY OUTCOMES:
postoperative pain and postoperative morphine consumption | postoperative 0 - 48 hours
  The effect of rectus sheath block on postoperative pain scores and morphine consumption in patients undergoing robotic prostatectomy will be investigated.

SECONDARY OUTCOMES:
urethral catheter pain | postoperative 0 - 48 hours
  The effect of rectus sheath block on urethral catheter pain in robotic prostatectomy operations will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Sami Kaan Coşarcan, Principal Investigator — American hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Amerikan Hastanesi, Istanbul
  - Koç Üniversitesi, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schiffmann J, Larcher A, Sun M, Tian Z, Berdugo J, Leva I, Widmer H, Lattouf JB, Zorn K, Haese A, Shariat SF, Saad F, Montorsi F, Graefen M, Karakiewicz PI. Differences in Patient Characteristics among Men Choosing Open or Robot-Assisted Radical Prostatectomy in Contemporary Practice - Analysis of Surveillance, Epidemiology, and End Results Database. Urol Int. 2017;98(1):40-48. doi: 10.1159/000447495. Epub 2016 Aug 4. PMID 27486887
- [Background] Woldu SL, Weinberg AC, Bergman A, Shapiro EY, Korets R, Motamedinia P, Badani KK. Pain and analgesic use after robot-assisted radical prostatectomy. J Endourol. 2014 May;28(5):544-8. doi: 10.1089/end.2013.0783. Epub 2014 Jan 30. PMID 24400824
- [Background] Desai N, El-Boghdadly K, Albrecht E. Epidural vs. transversus abdominis plane block for abdominal surgery - a systematic review, meta-analysis and trial sequential analysis. Anaesthesia. 2021 Jan;76(1):101-117. doi: 10.1111/anae.15068. Epub 2020 May 8. PMID 32385856
- [Background] Tran DQ, Bravo D, Leurcharusmee P, Neal JM. Transversus Abdominis Plane Block: A Narrative Review. Anesthesiology. 2019 Nov;131(5):1166-1190. doi: 10.1097/ALN.0000000000002842. PMID 31283738
- [Background] Chiancone F, Fabiano M, Ferraiuolo M, de Rosa L, Prisco E, Fedelini M, Meccariello C, Visciola G, Fedelini P. Clinical implications of transversus abdominis plane block (TAP-block) for robot assisted laparoscopic radical prostatectomy: A single-institute analysis. Urologia. 2021 Feb;88(1):25-29. doi: 10.1177/0391560320957226. Epub 2020 Sep 18. PMID 32945234